CLINICAL TRIAL: NCT07404228
Title: Multidimensional Study Designed to Develop a Methodological Framework Based on MRI Data to Predict Pathological Complete Response (pCR) in Patients With Locally Advanced Rectal Cancer After Neoadjuvant Treatment
Acronym: RESTAGE
Status: Not yet recruiting | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: PROICM 2025-07 RES
Record Dates: First submitted 2026-02-02; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Rectal Cancer; Chemoradiotherapy; Mri
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase 1 (Preclinical): An ex-vivo analysis of surgical specimens: 15 surgical specimens will be collected after surgery following neoadjuvant treatment. They will be imaged using a 3T MRI with advanced sequences, then returned to the pathology department. This ex vivo MRI will not affect sample preparation or preservation. MRI images will be aligned with histological sections using non-linear registration to compare MRI parameters with digital pathology data. This step will help identify MRI biomarkers that differentiate healthy tissue, post-treatment fibrotic tissue, and residual tumor. We will assess whether diffusion MRI and relaxometry measurements can predict pathological outcomes by analyzing parameters such as fractional anisotropy, mean diffusivity, and kurtosis, using surgical pathological information when available
- Phase 2 (Clinical): An in-vivo clinical MRI study.: The same advanced sequences will be added to MRIs performed during routine clinical care: the initial staging MRI before neoadjuvant chemoradiotherapy, the restaging MRI after treatment completion, and follow-up MRIs for patients managed with a non-operative Watch-and-Wait strategy. For each patient, we will collect imaging data, demographics, medical history, tumor characteristics, treatment details, pathology reports, and clinical follow-up (endoscopy and MRI). All data will be pseudonymized. The second phase involves developing a computational model to predict response to neoadjuvant therapy. A machine learning tool will be designed to predict complete pathological response based on quantitative MRI, standard clinical MRI, and clinical information
  Interventions: Other: questionnaire completion

INTERVENTIONS:
Other: questionnaire completion — For all patients, questionnaires will be completed:
  * At the MRI staging if applicable,
  * At the MRI restaging,
  * Every 3 months during the first year; and
  * Every 6 months during the second year.
  The following validated questionnaires will be used:
  * EORTC QLQ-C30 (overall quality of life)
  * EORTC QLQ-CR29 (colorectal cancer-specific symptoms)
  * EORTC IN-PATSAT32 (patient satisfaction with care)
  Groups: Phase 2 (Clinical): An in-vivo clinical MRI study.

SUMMARY:
Rectal cancer presents a significant global health challenge. Despite improvements in clinical outcomes, significant disparities persist across Europe. These differences are explained not only by the heterogeneity of risk factors and screening strategies, but also by variations in diagnostic and therapeutic approaches, which are highly dependent on medical imaging.

Standard treatment for locally advanced rectal cancer based on staging MRI is neoadjuvant treatment (NAT), for tumour downsizing and downstaging, followed by total mesorectal excision. In a significant proportion of cases, radical surgery leads to substantial long-term complications like sexual and urinary dysfunction, fecal incontinence, and impairment in daily activities. Given that up to 42% of patients show complete tumor regression at pathology (i.e. pathological complete response pCR), to avoid unnecessary radical surgery, non-operative management has become an attractive alternative when there are no signs of viable tumour after NAT (i.e. clinical complete response cCR). Such patients are candidates for Watch-and-Wait (W&W), an established active surveillance policy in specialized centers worldwide relying on clinical examination, endoscopy and MRI.

On the other hand, W&W carries a risk of local regrowth (persistence of microscopic residual disease despite apparent cCR). Even in expert hands, assessment of tumor response is not perfect and local regrowth based on current selection methods occurs in ~30% of cases. Although deferred surgery is a successful treatment with no apparent negative impact on local disease control, an increased rate of distant metastases has been recently reported.

Therefore, there is a critical unmet clinical need to detect complete responses after NAT and avoid unnecessary surgery with its associated morbidity and quality of life impairment risks, while also improving sensitivity for residual microscopic disease that will result in local regrowth and associated reduced disease-free survival.

Rectal cancer poses a burden not only on healthcare systems, but also on patient well-being. Patients frequently suffer from feelings of isolation and helplessness when faced with unpredicted disease-related situations, given the common difficulties to access high quality information and communicate with attending physicians. As such, there is a clear need to unburden healthcare facilities from unnecessary hospital visits, while improving patient outcomes, engagement, support and care.

ELIGIBILITY:
Inclusion Criteria for the preclinical phase :

* Age ≥18 years old;
* Have a confirmed diagnosis of locally advanced rectal cancer;
* Have completed neoadjuvant chemoradiotherapy;
* Be a candidate for surgical treatment with total mesorectal excision;
* Be willing and able to provide written informed consent;
* Affiliation to the French Social Security System.

Inclusion criteria for the clinical phase:

* Age ≥18 years old;
* Have a confirmed diagnosis of locally advanced rectal cancer;
* Require neoadjuvant chemoradiotherapy or have completed neoadjuvant chemoradiotherapy;
* Requires either surgical treatment or a non-surgical strategy ("Watch-and-Wait") after neoadjuvant chemoradiotherapy;
* Be willing and able to provide written informed consent;
* Affiliation to the French Social Security System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Preclinical phase: For patients requiring surgery after neoadjuvant chemoradiotherapy, a surgical consultation will be scheduled as part of routine care. The study will be explained, and an information sheet provided. Participation requires signing the informed consent by the patient and the investigating surgeon.
  Clinical phase: When a patient requires an MRI as part of their standard care, the study will be presented during the radiology consultation with an information sheet. If the patient agrees to participate, the informed consent form must be signed by the patient and the investigating physician.
  Patients may be included in the study at two possible times: during the MRI performed before neoadjuvant treatment (MRI staging), or during the re-evaluation MRI after neoadjuvant treatment (MRI restaging).
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
developpement and validation of a methodological framework based on advanced MRI data to predict pathological complete response in patients with locally advanced rectal cancer after neoadjuvant treatment | From the baseline to the end of follow up, assessed up to 27 months
  using the area under the ROC curve (AUC) to distinguish pathological complete response (pCR) from residual disease.

SECONDARY OUTCOMES:
evaluation of the overall diagnostic performance of the predictive model. | From the baseline to the end of follow up, assessed up to 27 months
  The overall diagnostic performance of the model will be evaluated using various indicators: Diagnostic accuracy: defined as the overall proportion of correct classifications, Sensitivity, Specificity, Positive predictive value and Negative predictive value
identification and validation of new MRI biomarkers capable of distinguishing residual tumor from benign fibrotic tissue, using ex vivo MRI of surgical specimens with direct correlation to histological data. | From the baseline to the end of follow up, assessed up to 27 months
  MRI-histology correlation: statistical correlation between advanced MRI data (derived from ex vivo acquisitions) and the corresponding histological measurements of surgical specimens. Regions of interest (ROIs) defined on ex vivo MRI will be matched with digitized histology. This criterion will validate the new biomarkers.
establishment of a rectal MRI database to support this project and future research. | From the baseline to the end of follow up, assessed up to 27 months
  Establishment of a data registry: creation of a functional, populated database of rectal cancer cases that is compliant with the FAIR principles (Findable, Accessible, Interoperable, Reusable).
assessment of the impact of the disease and therapeutic strategies on patients' quality of life. | From the baseline to the end of follow up, assessed up to 27 months
  Quality of life scores: scores obtained from standardized questionnaires collected via a digital application to assess the overall impact of the disease and treatments on patients' lives. These will be analyzed using linear mixed models, comparing the surgical group with the "Watch-and-Wait" group over time.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie NOUGARET, PHD, Study Director — ICM Co. Ltd.
Locations (1):
- ICM, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients All participant data collected during the trial, after encoding with an inclusion number, 1st letter of the name and surname may be shared.
  The data of the participants will be available upon request and with the completion of a contract between the promoter and the applicant.
  The study protocol, the statistical analysis plan (PAS) and the analytical code may also be subject to data sharing as part of a transfer contract (RGPD)

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Heald RJ, Ryall RD. Recurrence and survival after total mesorectal excision for rectal cancer. Lancet. 1986 Jun 28;1(8496):1479-82. doi: 10.1016/s0140-6736(86)91510-2. PMID 2425199
- [Background] Wrenn SM, Cepeda-Benito A, Ramos-Valadez DI, Cataldo PA. Patient Perceptions and Quality of Life After Colon and Rectal Surgery: What Do Patients Really Want? Dis Colon Rectum. 2018 Aug;61(8):971-978. doi: 10.1097/DCR.0000000000001078. PMID 29944576
- [Background] Maas M, Nelemans PJ, Valentini V, Das P, Rodel C, Kuo LJ, Calvo FA, Garcia-Aguilar J, Glynne-Jones R, Haustermans K, Mohiuddin M, Pucciarelli S, Small W Jr, Suarez J, Theodoropoulos G, Biondo S, Beets-Tan RG, Beets GL. Long-term outcome in patients with a pathological complete response after chemoradiation for rectal cancer: a pooled analysis of individual patient data. Lancet Oncol. 2010 Sep;11(9):835-44. doi: 10.1016/S1470-2045(10)70172-8. Epub 2010 Aug 6. PMID 20692872
- [Background] Garcia-Aguilar J, Shi Q, Thomas CR Jr, Chan E, Cataldo P, Marcet J, Medich D, Pigazzi A, Oommen S, Posner MC. A phase II trial of neoadjuvant chemoradiation and local excision for T2N0 rectal cancer: preliminary results of the ACOSOG Z6041 trial. Ann Surg Oncol. 2012 Feb;19(2):384-91. doi: 10.1245/s10434-011-1933-7. Epub 2011 Jul 14. PMID 21755378
- [Background] Park IJ, Yu CS. Current issues in locally advanced colorectal cancer treated by preoperative chemoradiotherapy. World J Gastroenterol. 2014 Feb 28;20(8):2023-9. doi: 10.3748/wjg.v20.i8.2023. PMID 24587677
- [Background] Dattani M, Heald RJ, Goussous G, Broadhurst J, Sao Juliao GP, Habr-Gama A, Perez RO, Moran BJ. Oncological and Survival Outcomes in Watch and Wait Patients With a Clinical Complete Response After Neoadjuvant Chemoradiotherapy for Rectal Cancer: A Systematic Review and Pooled Analysis. Ann Surg. 2018 Dec;268(6):955-967. doi: 10.1097/SLA.0000000000002761. PMID 29746338
- [Background] Sao Juliao GP, Habr-Gama A, Vailati BB, Perez RO. The good, the bad and the ugly: rectal cancers in the twenty-first century. Tech Coloproctol. 2017 Jul;21(7):573-575. doi: 10.1007/s10151-017-1651-7. Epub 2017 Jun 19. No abstract available. PMID 28631136
- [Background] Beets-Tan RGH, Lambregts DMJ, Maas M, Bipat S, Barbaro B, Curvo-Semedo L, Fenlon HM, Gollub MJ, Gourtsoyianni S, Halligan S, Hoeffel C, Kim SH, Laghi A, Maier A, Rafaelsen SR, Stoker J, Taylor SA, Torkzad MR, Blomqvist L. Magnetic resonance imaging for clinical management of rectal cancer: Updated recommendations from the 2016 European Society of Gastrointestinal and Abdominal Radiology (ESGAR) consensus meeting. Eur Radiol. 2018 Apr;28(4):1465-1475. doi: 10.1007/s00330-017-5026-2. Epub 2017 Oct 17. PMID 29043428
- [Background] Socha J, Kepka L, Michalski W, Paciorek K, Bujko K. The risk of distant metastases in rectal cancer managed by a watch-and-wait strategy - A systematic review and meta-analysis. Radiother Oncol. 2020 Mar;144:1-6. doi: 10.1016/j.radonc.2019.10.009. Epub 2019 Nov 8. PMID 31710938
- [Background] van der Valk MJM, Hilling DE, Bastiaannet E, Meershoek-Klein Kranenbarg E, Beets GL, Figueiredo NL, Habr-Gama A, Perez RO, Renehan AG, van de Velde CJH; IWWD Consortium. Long-term outcomes of clinical complete responders after neoadjuvant treatment for rectal cancer in the International Watch & Wait Database (IWWD): an international multicentre registry study. Lancet. 2018 Jun 23;391(10139):2537-2545. doi: 10.1016/S0140-6736(18)31078-X. PMID 29976470
- [Background] Nasir I, Fernandez L, Vieira P, Pares O, Santiago I, Castillo-Martin M, Domingos H, Cunha JF, Carvalho C, Heald RJ, Beets GL, Parvaiz A, Figueiredo N. Salvage surgery for local regrowths in Watch & Wait - Are we harming our patients by deferring the surgery? Eur J Surg Oncol. 2019 Sep;45(9):1559-1566. doi: 10.1016/j.ejso.2019.04.006. Epub 2019 Apr 13. PMID 31006589
- [Background] Fernandez LM, Sao Juliao GP, Renehan AG, Beets GL, Papoila AL, Vailati BB, Bahadoer RR, Kranenbarg EM, Roodvoets AGH, Figueiredo NL, Van De Velde CJH, Habr-Gama A, Perez RO; International Watch & Wait Database (IWWD) Consortium. The Risk of Distant Metastases in Patients With Clinical Complete Response Managed by Watch and Wait After Neoadjuvant Therapy for Rectal Cancer: The Influence of Local Regrowth in the International Watch and Wait Database. Dis Colon Rectum. 2023 Jan 1;66(1):41-49. doi: 10.1097/DCR.0000000000002494. Epub 2022 Oct 21. PMID 36515514
- [Background] Smith JJ, Strombom P, Chow OS, Roxburgh CS, Lynn P, Eaton A, Widmar M, Ganesh K, Yaeger R, Cercek A, Weiser MR, Nash GM, Guillem JG, Temple LKF, Chalasani SB, Fuqua JL, Petkovska I, Wu AJ, Reyngold M, Vakiani E, Shia J, Segal NH, Smith JD, Crane C, Gollub MJ, Gonen M, Saltz LB, Garcia-Aguilar J, Paty PB. Assessment of a Watch-and-Wait Strategy for Rectal Cancer in Patients With a Complete Response After Neoadjuvant Therapy. JAMA Oncol. 2019 Apr 1;5(4):e185896. doi: 10.1001/jamaoncol.2018.5896. Epub 2019 Apr 11. PMID 30629084
- [Background] Tsunoda A, Nakao K, Hiratsuka K, Yasuda N, Shibusawa M, Kusano M. Anxiety, depression and quality of life in colorectal cancer patients. Int J Clin Oncol. 2005 Dec;10(6):411-7. doi: 10.1007/s10147-005-0524-7. PMID 16369745
- See also: Rectal cancer: ESMO clinical practice guidelines — https://www.esmo.org/guidelines/esmo-clinical-practice-guideline-localised-rectal-cancer